CLINICAL TRIAL: NCT00973635
Title: The Web-Based Education of Beginning Interns on Handoffs
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Diane Wayne, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: STU00009658
Record Dates: First submitted 2009-08-21; First posted 2009-09-09 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Medical Interns and Medical Students
Keywords: education; web-based intervention; patient care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional training (No Intervention): Patients of subjects with no detailed curriculum for handoff skills during non-intervention months.
  Learners provided a brief outline of how to perform discharge summaries (handout).
  Learners given two core articles describing some of the communication issues regarding handoff safety.
  Handoff teaching left to discretion of the subintern's team (typically the "see one, do one, teach one" method).
  No feedback given to these subinterns on their performance of their handoff skills.
- Intervention (Experimental): Group that receives educational intervention.
  Interventions: Other: Web-based education

INTERVENTIONS:
Other: Web-based education — Patients of subjects who were required to complete 10 web-based, independent learning modules. Each subject given a course packet which includes 13 required "core articles" pertaining to handoff skills. Each subject receives immediate feedback to each web-case with correct answers and suggested readings. Each subject given individualized feedback on their scores for summaries, instructions, and sign outs.
  Arms: Intervention

SUMMARY:
A handoff is defined as the transfer of role and responsibility from one person to another in a physical or mental process. Current evidence shows that handoffs between medical providers are both common, and fraught with potential for harm. In spite of these problems, handoff skills are rarely discussed or practiced. Currently, there are few curricula available in the literature regarding the teaching of handoff skills. The purpose of the investigators' study is to develop a curriculum focusing on key handoff safety issues. The investigators plan to create an independent learning tutorial that would be easily administered to all beginning interns (medical subinterns and 2nd month pgy1 medical interns), that would be accessible across multiple sites, that would increase learner knowledge regarding key handoff safety issues, and would improve trainee satisfaction with the handoff process. The investigators' goal is to make this curriculum practical and time efficient. The investigators' hope is that the educational intervention would also have a measurable impact on the quality of patient care.

DETAILED DESCRIPTION:
A handoff is defined as the transfer of role and responsibility from one person to another in a physical or mental process.1 Handoffs in some fields, like commercial aviation and professional athletics, are highly visible. In these situations, the handoff process is practiced repeatedly and near misses are reviewed to avoid future errors. In other professions, such as medicine, handoffs occur behind the scenes and the lack of public visibility can result in poor recognition of problems.

Current evidence shows that handoffs between medical providers are both common, and fraught with potential for harm. On the inpatient side, the scope of preventable medical errors became visible to the public in 1999 with the publication of "To Err is Human." The Institute of Medicine estimated that between 44,000 and 98,000 patients die each year in U.S. hospitals as a result of avoidable medical errors.2 Later studies estimated that communication failures among health care team members was the root cause of an estimated 75% of these hospital adverse events.3 Hospitalizations are complex and communication errors can occur at multiple points during a hospital stay. Miscommunication during patient care handoffs is a particular area of concern. Due to the sheer number of handoffs which occur, the potential for handoffs to cause harm is enormous. At one major U.S. academic medical center, 15 handoffs occurred per patient during a typical 5 day hospital stay and each intern on the medical service was involved in more than 300 handoffs over a 1-month rotation.4

While handoff errors occurring as an inpatient are certainly a problem, they may just be the tip of the error iceberg. Available data would suggest that adverse events related to poor handoffs at discharge are an even larger patient safety issue. In one small study, nearly 50% of hospitalized medical patients experienced at least 1 medical error after discharge relating to either medication continuity, diagnostic workup, or test follow-up issues.5 In a large prospective Canadian study, 23% of discharged patients experienced a significant adverse event within 5 weeks, and more than half of these adverse events were judged to be preventable.6 Many of these adverse events after discharge were "handoff errors" related to discontinuity of care and breakdown in the communication between patients, hospital physicians and outpatient primary care providers. A 2007 review article on the transfer of information between hospital-based physicians and primary care physicians confirmed that direct communication was rare between hospital physicians and primary care physicians, summaries were often poor quality, and the availability of discharge summaries was low at initial outpatient follow-up visits. The study investigators estimated that missing discharge summaries negatively affected 25% of patients.7

In spite of these communication deficits, handoff skills are rarely discussed or practiced. Formal instruction on handoff skills is lacking at many US medical schools, in fact a survey of clerkship directors in 2004 found that only 8% of schools had any curriculum on handoffs.1,8 In most academic medical centers, beginning interns (new pgy1 interns and m4 subinterns) are responsible for performing the majority of handoffs4 (inpatient night float handoffs, team-to-team transfer handoffs, outpatient discharge handoffs, and others) in spite of evidence suggesting that interns are more likely to commit handoff errors.9 In lieu of formal training, beginning interns often learn their handoff techniques using the infamous "see one, do one, teach one" method. However, this is not the optimal format for adult learners acquiring a new skill.10 There is a perception among many hospital physicians that patients are "sicker and discharged quicker" than ever before.11 Without formal education, beginning interns may not have the skills required to perform these complex handoffs safely and effectively.

Currently, there are few curricula available in the literature regarding the teaching of handoff skills. One single-institution study exists regarding the teaching of discharge summary skills.12 This study confirmed discharge summary quality can be improved with a targeted educational intervention, but the intervention was based on recurring faculty-delivered lectures and would not be easily implemented across multiple sites without investing in significant faculty development programs. Another single-institution study described the development of a curriculum on verbal sign out skills, but again, this intervention required noon conference participation and was only able to capture one-quarter of the targeted housestaff due to scheduling issues and patient care conflicts.4 Because of the faculty training involved, the hands-on time needed, and the difficulty of scheduling educational conferences for house officers already struggling with work-hours restrictions; it would be difficult to deliver these face-to-face programs on a large scale and ensure that all trainees receive the interventions.

The purpose of study is to develop a curriculum focusing on key handoff safety issues. The investigators plan to create an independent learning tutorial that would be easily administered to all beginning interns (medical subinterns and 2nd month pgy1 medical interns), that would be accessible across multiple sites, that would increase learner knowledge regarding 25 key handoff safety issues, and would improve trainee satisfaction with the handoff process. The study's goal is to make this curriculum practical and time efficient. The investigators hope is that the educational intervention would also have a measurable impact on the quality of patient care.

ELIGIBILITY:
Inclusion Criteria:

* All discharged patients of Sub-interns and Interns

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Measurement of the quality of three discharge summaries, selected at random, using standardized content scoring card | up to 1 year after study

SECONDARY OUTCOMES:
re-admission rates and determination of preventability for each re-admission case | 1 year